CLINICAL TRIAL: NCT03858543
Title: Fractional Laser Assisted Delivery of Sculptra® for the Treatment of Striae: FADeS Trial
Brief Title: Fractional Laser Assisted Delivery of Sculptra® for the Treatment of Striae
Acronym: FADeS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Principal Investigator, aamir siddiqui, Division Head - Plastic & Reconstruction Surgery, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11951
Record Dates: First submitted 2019-02-18; First posted 2019-02-28 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Striae Distensae
Keywords: Stretch marks; Fractional laser therapy; Poly-L lactic acid; Sculptra
MeSH Terms: conditions — Striae Distensae | interventions — New-Fill

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Fractional laser treatment & Poly-L Lactic Acid (Sculptra) (Experimental): One Fractional laser treatment on half of the body with Sciton Laser and Scluptra
  Interventions: Drug: Poly-L Lactic Acid; Device: Fractional laser treatment
- Fractional laser treatment (Active Comparator): One Fractional laser treatment on half of the body with Sciton Laser
  Interventions: Device: Fractional laser treatment

INTERVENTIONS:
Drug: Poly-L Lactic Acid — After initial treatment, reassessment will be conducted at 3 follow-up visits. Photographs will be taken for blinded evaluators to compare post-treatment to the original pre-treatment photographs. At final visit, a questionnaire will be administered to rate treatment satisfaction.
  Other Names: Sculptra
  Arms: Fractional laser treatment & Poly-L Lactic Acid (Sculptra)
Device: Fractional laser treatment — After initial treatment, reassessment will be conducted at 3 follow-up visits. Photographs will be taken for blinded evaluators to compare post-treatment to the original pre-treatment photographs. At final visit, a questionnaire will be administered to rate treatment satisfaction.
  Other Names: Sciton Laser

SUMMARY:
This study evaluates the efficacy of treatment of striae distensae using the combined modality of fractional laser and poly-L lactic acid (Sculptra).

DETAILED DESCRIPTION:
Striae Distensae (SD) is a form of scarring that can oftentimes be quite disfiguring and emotionally distressing to individuals.

Fractional laser therapy has been used by doctors to treat stretch marks by stimulating collagen growth.

Poly-L lactic acid also promotes collagen growth in the areas injected.

The combination of laser and poly-L lactic acid might provide the optimal treatment modality for SD by decreasing the appearance of atrophic scars.

ELIGIBILITY:
Inclusion Criteria:

* Subject has bilateral striae alba
* Subject has stable body weight for at least 6 months with Fitzpatrick skin type 1-4

Exclusion Criteria:

* Subject has striae rubra
* Pregnant
* History of adverse effects to phototherapy
* Subject has single sided lesions
* Subject has immunosuppression
* Subject has radiation therapy to the study area
* Subject has topical or oral steroid use or chemotherapy within the last 6 months
* History of keloids or hypertrophic scar

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Stretch Mark Size | Baseline (Pre-treatment) vs. 3 Months, 4 Months, 5 Months, 6 Months
  Modified Manchester Scar Scale was used to assess stretch mark reduction compared to pre-treatment photographs. The range of each subscale is between 4-26. A higher value represents a worse outcome. A value of 26 is the maximum score and represents the worst outcome. A value of 4 is the minimum score and represents the best outcome. Subscales are then summed to compute a total score.

SECONDARY OUTCOMES:
Treatments Superiority Assessment | 3 Months
  Modified Manchester Scar Scale was used to assess and judge whether erbium-YAG fractionated laser therapy plus Sculptra is superior to laser therapy alone. The range of each subscale is between 4-26. A higher value represents a worse outcome. A value of 26 is the maximum score and represents the worst outcome. A value of 4 is the minimum score and represents the best outcome. Subscales are then summed to compute a total score.
Treatments Superiority Assessment | 4 Months
  Modified Manchester Scar Scale was used to assess and judge whether erbium-YAG fractionated laser therapy plus Sculptra is superior to laser therapy alone. The range of each subscale is between 4-26. A higher value represents a worse outcome. A value of 26 is the maximum score and represents the worst outcome. A value of 4 is the minimum score and represents the best outcome. Subscales are then summed to compute a total score.
Treatments Superiority Assessment | 5 Months
  Modified Manchester Scar Scale was used to assess and judge whether erbium-YAG fractionated laser therapy plus Sculptra is superior to laser therapy alone. The range of each subscale is between 4-26. A higher value represents a worse outcome. A value of 26 is the maximum score and represents the worst outcome. A value of 4 is the minimum score and represents the best outcome. Subscales are then summed to compute a total score.
Treatments Superiority Assessment | 6 Months
  Modified Manchester Scar Scale was used to assess and judge whether erbium-YAG fractionated laser therapy plus Sculptra is superior to laser therapy alone. The range of each subscale is between 4-26. A higher value represents a worse outcome. A value of 26 is the maximum score and represents the worst outcome. A value of 4 is the minimum score and represents the best outcome. Subscales are then summed to compute a total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States